CLINICAL TRIAL: NCT04867772
Title: COmmunity Based Rehabilitation After Knee Arthroplasty (CORKA): A Prospective Two Arm Individually Randomised Controlled Trial
Brief Title: Community Based Rehabilitation After Knee Arthroplasty
Acronym: CORKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: HTA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3.0 25Nov2015
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Knee Arthroplasty

STUDY DESIGN:
Intervention Model Description: 2 arm RCT
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Other): Participants will receive the care that would usually be received in the local hospital setting. this has been determined as between 1 and 6 sessions of physiotherapy
  Interventions: Other: Home based rehabilitation
- Intervention (Experimental): Participants will receive a home based rehabilitation programme with 1-7 sessions of physiotherapy delivered over 12 weeks.
  Interventions: Other: Home based rehabilitation

INTERVENTIONS:
Other: Home based rehabilitation

SUMMARY:
Background The CORKA study was developed in response to a commissioned call by the National Institute for Health Research (NIHR) Health Technology Assessment (HTA) programme for research into a functional home based rehabilitation programme for patients who may be at risk of poor outcome after knee arthroplasty.

Design The CORKA trial is a prospective individually randomised controlled trial with blinded outcome assessment at baseline, 6 and 12 months. The study will also include a qualitative and a health economic analysis. Participants will be randomised to one of two arms, 'home-based rehabilitation' or 'Usual Care'. Those in the usual care arm will receive a minimum of 1 and a maximum of 6 sessions of physiotherapy as delivered locally, e.g. class, one to one, etc. Those in the intervention arm will receive 7 sessions of a functional rehabilitation programme over a 12 week timescale. The intervention will be delivered using physiotherapists and physiotherapy assistants in the participants' home. Participants will be followed up at 6 months and 12 months

ELIGIBILITY:
Inclusion Criteria:

Participant is willing and able to give informed consent for participation in the study Male or Female, aged 55 years or above Primary unilateral KR as a scheduled procedure Deemed by study screening tool developed to be at risk of poor outcome Happy to allow physiotherapy teams to attend their home to deliver the Community based rehabilitation programme if randomised to the intervention arm.

Exclusion Criteria:

Any absolute contraindications to exercise Severe cardiovascular or pulmonary disease (New York Heart Association III-IV) Severe dementia, assessed using the hospital dementia screening tool Rheumatoid arthritis Further lower limb arthroplasty surgery planned within 12 months. Serious perioperative complications

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
To compare the patient reported functional outcome and quality of life of the CORKA trial rehabilitation protocol versus standard care in participants at risk of poor outcome after knee replacement | over 12 months
  functional outcome LLFDI

SECONDARY OUTCOMES:
To assess the safety and serious adverse events associated with the treatment programme: SAE | over 12 months
  Safe and effective SAE reports
To assess the acceptability to the treatment programme for patients and therapists through both a RCT and a nested qualitative study | over 12 months
  Qualatative interviews
To assess the cost effectiveness of the different treatment strategies | over 12 months
  QALY